CLINICAL TRIAL: NCT02973217
Title: Prospective, Open, Non Comparative Trial to Evaluate Safety and Feasibility of Immunostimulating Interstitial Laser Thermotherapy (imILT) in Stage III Pancreatic Carcinoma
Brief Title: Immunostimulating Interstitial Laser Thermotherapy in Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Laserthermia Systems AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-2015-008
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Neoplasms Pancreatic
Keywords: Hyperthermia, Induced; Laser Coagulation; Laser Therapy
MeSH Terms: conditions — Pancreatic Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- imILT (Experimental): Immunostimulating Interstitial Laser Thermotherapy (imILT)
  Interventions: Device: Immunostimulating Interstitial Laser Thermotherapy

INTERVENTIONS:
Device: Immunostimulating Interstitial Laser Thermotherapy

SUMMARY:
Thermotherapy is a technology aiming at destroying tissue, for example tumor tissue. Immunostimulating Interstitial Laser Thermotherapy (imILT) is a specific form of thermotherapy, which, in addition to destroying tumor tissue, has been optimized to cause a tumor specific immunologic response. In laboratory animals the imILT method has also been shown to induce a so called abscopal effect. This means that when one tumor is treated with imILT other, untreated, tumors also decrease in size.

The purpose of this trial is to evaluate efficiency when it comes to local tumor destruction of the imILT treatment method in patients diagnosed with pancreatic cancer. The purpose is also to investigate the functionality and safety as well as understanding of the subsequent immunological effects.

This trial is prospective, open and non-randomized. Five patients diagnosed with pancreatic cancer will be treated in this trial, which is estimated to be carried out during a time period of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Cytohistological diagnosis of ductal pancreatic adenocarcinoma .
* Stage III disease (see above).
* The patient is not a candidate for continued chemotherapy or (chemo)radiotherapy due to lack of demonstrable efficiency or to the side effects of the drugs.
* Age between 18 and 80 years.
* Anticipated compliance with treatment and follow-up.
* Double informed consent for both imILT and possible surgery with radical intent (in the event of pre-operative overstaging).
* At least a part of the tumor can be treated with imILT without damage to surrounding vital structures.
* Have an ECOG performance status < 1 (l'Eastern Cooperative Oncology Group)

Exclusion Criteria:

* Not a candidate for laparotomy.
* Becoming resectable after neoadjuvant chemotherapy.
* Other simultaneous treatments for the same neoplasm.
* Simultaneous other malignancies except for basal cell carcinoma.
* HIV positive.
* Active autoimmune disease.
* Systemic corticosteroid medication.
* Pregnancy or nursing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) | 36 months
  Evaluation of adverse events.

SECONDARY OUTCOMES:
Inflammatory response in circulation measured by quantification of inflammatory cell populations | 36 months
  Quantification of cellular infiltrate and activation markers by flow cytometry.
Disease progression | 36 months
  Analysis of the percentage of patients with no new oncological events.
Evaluation of Quality of Life (using questionnaires) | 36 months
  Evaluation of Quality of Life is evaluated using standardized questionnaires.
Usability of the device as evaluated by treatment logs | 36 months
  Evaluation of the laser system by analysis of treatment logs of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut J. Paoli et L. Calmettes (IPC), Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paiella S, Casetti L, Ewald J, Marchese U, D'Onofrio M, Garnier J, Landoni L, Gilabert M, Manzini G, Esposito A, Secchettin E, Malleo G, Lionetto G, De Pastena M, Bassi C, Delpero JR, Salvia R, Turrini O. Laser Treatment of Pancreatic Cancer with Immunostimulating Interstitial Laser Thermotherapy Protocol: Safety and Feasibility Results From Two Phase 2a Studies. J Surg Res. 2021 Mar;259:1-7. doi: 10.1016/j.jss.2020.10.027. Epub 2020 Dec 2. PMID 33278792